CLINICAL TRIAL: NCT02559479
Title: A Study to Assess the Effect of a Normal vs. High Protein Diets in Carbohydrates Metabolism in Obese Subjects With Diabetes or Prediabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Aragones de Ciencias de la Salud (Other Government)
Responsible Party: Principal Investigator, Fernando Civeira, Professor, Instituto Aragones de Ciencias de la Salud
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEICA;PI/15/0183
Record Dates: First submitted 2015-09-22; First posted 2015-09-24 (Estimated); Last update posted 2016-12-02 (Estimated); Status verified 2016-12

CONDITIONS: Weight Loss; Obesity; Diabetes; Diet, Reducing; Carbohydrates; Protein
MeSH Terms: conditions — Weight Loss; Obesity; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 18%-Protein diet (Active Comparator): Energy-restricted diet wit the following composition: 18% protein, 30% fat and 52% carbohydrates
  Interventions: Behavioral: Weight loss interventional study with a low-calorie 18%-protein diet
- 35%-Protein diet (Active Comparator): Energy-restricted diet wit the following composition: 35% protein, 30% fat and 35% carbohydrates
  Interventions: Behavioral: Weight loss interventional study with a low-calorie 35%-protein diet

INTERVENTIONS:
Behavioral: Weight loss interventional study with a low-calorie 18%-protein diet
  Arms: 18%-Protein diet
Behavioral: Weight loss interventional study with a low-calorie 35%-protein diet
  Arms: 35%-Protein diet

SUMMARY:
The objective of the study is to assess the effect of low-calorie diets with normal (18%) vs. high (35%) protein (mainly coming from animal source) composition on body weight and carbohydrates metabolism in overweight and obese subjects with pre-diabetes or diabetes. A dietary intervention is carried out during 6 months in 100 subjects who are individually randomized to an energy-restricted diet with two types of macronutrients composition: 1) 35% protein, 30% fat and 35% carbohydrates and 2) 18% protein, 30% fat and 52% carbohydrates. Around 80% of total protein in diet comes from animal source (of whom around 40% from lean red meat). Subjects are provided with weekly menus and different recipes to use them as part of the diet. Monitoring visits with the nutritionist will be performed every 15 days. At the beginning of the study, after 3 and 6 months, the following parameters are determined: anthropometric (weight, waist circumference, body mass index and body composition), blood pressure, dietary (72-hours dietary registry) and exercise and biochemical analysis (total cholesterol, triglycerides, HDL cholesterol, LDL cholesterol, apolipoproteins A1 and B, iron, transferring, ferritin, uric acid, glucose, HbA1c, insulin, adiponectin and resistin). Urine samples are also collected to assess microalbuminuria and ureic nitrogen.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-70 years old.
* Body mass index between 27.5 - 40.
* Steady weight (± 4 kg) in the last 2 months.
* Glycated hemoglobin between 6 - 7%.

Exclusion Criteria:

* Anti-diabetic drugs (oral or subcutaneous) in the last 2 months.
* Lipid-lowering drugs in the last 2 months.
* Gouty arthritis in the last 2 years or uric acid > 735 mg/dl.
* Presence of uncontrolled endocrinological pathology (including hypothyroidism).
* Hepatic chronic disease (glomerular filtration rate < 45 ml/min).
* Renal, inflammatory or tumoral diseases.
* Drugs which could interfere in glucose or lipid metabolism such as androgens, corticosteroids (except for those with topic administration) and estrogen replacement therapy.
* Intake of functional foods with plant sterols in the past 6 weeks.
* High alcohol intake (> 30 g per day).
* Any serious disease which involves less than 1 year life expectancy or, in investigators judgment, limit the follow-up of an homogeneous diet throughout the study.
* Pregnancy or intention of pregnancy during the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-09; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Change in glucose. | After 3 and 6 months of intervention.
Change in glycated hemoglobin. | After 3 and 6 months of intervention.
Change in insulin resistance (HOMA index). | After 3 and 6 months of intervention.

SECONDARY OUTCOMES:
Change in body weight. | After 3 and 6 months of intervention.
Change in body composition. | After 3 and 6 months of intervention.
Change in waist circumference. | After 3 and 6 months of intervention.
Change in lipid profile (total cholesterol, LDL cholesterol, HDL cholesterol, non HDL cholesterol, triglycerides and apolipoproteins). | After 3 and 6 months of intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Civeira, MD, PhD, Principal Investigator — Unidad Clínica y de Investigación en Lípidos y Arteriosclerosis; Hospital U. Miguel Servet; IIS Aragón
Locations (1):
- Fernando Civeira, Zaragoza, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Marco-Benedi V, Perez-Calahorra S, Bea AM, Lamiquiz-Moneo I, Baila-Rueda L, Cenarro A, Civeira F, Mateo-Gallego R. High-protein energy-restricted diets induce greater improvement in glucose homeostasis but not in adipokines comparing to standard-protein diets in early-onset diabetic adults with overweight or obesity. Clin Nutr. 2020 May;39(5):1354-1363. doi: 10.1016/j.clnu.2019.06.005. Epub 2019 Jun 15. PMID 31255349